CLINICAL TRIAL: NCT03923608
Title: Localized Muscle Resistance Test: Identification and Use of Parameters for Prescription of Exercise Resisted in Different Evaluation Tools
Brief Title: Reliability of a Endurance and a Strength Test for Shoulder Rotation
Status: Completed | Type: Observational
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Jéssica Kirsch Michelleti, Principal Investigator, São Paulo State University
Other Study IDs: SP-Unesp
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- strength test: The maximum strength test of external shoulder rotators will be performed on 5 different tools with specific protocols.
  Interventions: Diagnostic Test: Maximal muscle strength Test
- Endurance test: Test designed by the Laboratory of Sports Physical Therapy (LAFIDE) of FCT / UNESP - Presidente Prudente, used in the prescription of training for gain of localized muscular endurance. Will be realized in the tools: Isokinetic dynamometer, elastic bands, pulley and halter.
  The test will consist of the maximum possible repetitions (until fatigue) with loads of 70%, 80% and 90% of the maximum force (in different sessions).
  Interventions: Diagnostic Test: Exhaustion test

INTERVENTIONS:
Diagnostic Test: Maximal muscle strength Test — 1RM test performed in 5 different tools (Elastic Band, Pulley, halter, digital dynamometer and isokinetic dynamometer)
  Groups: strength test
Diagnostic Test: Exhaustion test — Test performed until individual exhaustion in 5 different tools (Elastic Band, Pulley, halter and isokinetic dynamometer)
  Groups: Endurance test

SUMMARY:
Introduction: Verification of the progression of individuals submitted to training programs is performed by diagnostic tests with a focus on strength and muscular endurance. Among the tools used are the elastic bands, the halter, the pulley, the digital dynamometer and, additionally, the isokinetic dynamometer, considered the gold standard of evaluation. However, there is a lack of standardization in assessments and scarcity in the exploration of some tools and some muscle groups. Observation is often restricted to a particular study design and makes comparisons difficult even with the use of the same tool. Thus, to include different clinical possibilities in the same scenario can enrich the discussion about the topic. Objective: To develop and analyze the validity and reliability of a maximal muscle strength test for the external rotator muscles of the shoulder in five tools; To develop and analyze the validity and reliability of a localized resistance test for the external rotator muscles of shoulder in three different percentages of maximum strength (60%, 70%, 80%) in four tools; To characterize by means of the physiological response the localized muscular endurance test with the load that presents with the highest reliability values in each tool. Method: The study will consist of a sample of 50 participants of both genders, and will be performed in 3 steps: (1) Validation and reliability of the maximum muscle strength test; (2) Reliability of the muscular endurance test (MET); (3) Physiological characterization of the muscular endurance test (MET). Stage 1 will be held in 3 sessions (familiarization, test and retest) in which participants will perform 5 tests of maximum strength with different tools (elastic bands, pulley, halter, digital dynamometer and isokinetic dynamometer). Stage 2, consisting of 6 sessions, will be tested and retest of a muscular endurance test with different loads (70%, 80% and 90% of maximum force) with the same devices of step 1, except the digital dynamometer. In Step 3 participants will be selected with the lowest variations between the test and retest in the variable "time" to perform the physiological characterization of the test with the different tools. In order to observe the physiological response, we will analyze the lactic anaerobic (lactate concentration), allelic anaerobic (post-exercise oxygen uptake (EPOC) and aerobic (VO 2 values) parameters). The statistical package SPSS Statistics 22.0 will be used to conduct the analyzes. Key words: Fatigue, Physical resistance, Muscle strength, Lactate.

ELIGIBILITY:
Inclusion Criteria: should report the absence of:

* anemia,
* diabetes,
* cardiovascular disease,
* and upper limb and spinal muscular injuries in the last six months

Exclusion Criteria:

* absence at any study session and
* episode of muscle-tendon or osteoarticular injury in the upper limbs during the study.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample is composed of apparently healthy young men, of both genders, between 13 and 30 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Maximal force (kilograms) | Stage 1 - 0 minutes after strength test
  The maximum force of the participant shall be measured with the values presented in kilogram
Time (seconds) | Stage 2 - 0 minutes after Endurance test
Number of repetitions | Stage 2 -0 minutes after Endurance test
Anthropometric evaluation | Stage 1 - 10 minutes before stregth test
  To determine the value corresponding to the body mass, the volunteers will be evaluated by a digital scale (Tanita BC554, Iron Man / Inner Scaner - Tanita, Illinois, United States). Stature values will be obtained by means of a stadiometer (Sanny - American Medical do Brasil, São Paulo, Brazil). From these values it will be possible to calculate the Body Mass Index (BMI), determined by the ratio of weight to height squared.
Psychological Questionnaire | Stage 1 - 10 minutes before stregth test
  The questionnaire aims to subjectively document physical and metal readiness scores for exercise, fatigue, vigor, drowsiness, and muscle pain. Participants will be instructed to mark a dash on a visual analogue scale of 10 centimeters between two extremes, zero being "least possible" and 10 indicating "most possible" for each classification60. This questionnaire will be applied at the beginning of all sessions.
International Physical Activity Questionnaire (IPAQ) | Stage 1 - 10 minutes before stregth test
  The IPAQ questionnaire is an instrument developed to estimate the level of habitual practice of physical activity. Sedentary - Does not perform any physical activity for at least 10 continuous minutes; Insufficiently Active - Individuals who engage in physical activity for at least 10 continuous minutes per week, but insufficiently to be classified as active. A) Perform 10 continuous minutes of physical activity, following at least one of the following criteria: frequency - 5 days/week or duration - 150 minutes/week; B) Does not meet any of the criteria of the recommendation cited in under-active individuals A; Active - a) vigorous physical activity - ≥ 3 days/week and ≥ 20 minutes/session; b) moderate or walking - ≥ 5 days/week and ≥ 30 minutes/session; c) any added activity: ≥ 5 day/week and ≥ 150 min/week; Very Active - a) vigorous - ≥ 5 days/week and ≥ 30 min/session; b) vigorous - ≥ 3 days/week and ≥ 20 min/session + moderate and or ≥ 5 days/week and ≥ 30 min/session.
Borg's Perception of Effort Scale | Stage 2 - 0 minutes after endurance test in all tools
  The degree of subjective effort reported by the participants in relation to the upper limbs will be analyzed using the Borg scale of perception of effort of 6 to 20 points, 6 corresponding to the "very easy" and 20 to "exhaustive".
Perceived effort | Stage 2 - 0 minutes after endurance test in all tools
  The perceived exertion of the resisted exercise will be evaluated through the OMNI Resistance Exercise Scale for Perceived Effort62,63, which consists of an ordinal scale of 0 to 10, 0 being extremely easy and 10 extremely difficult.
Recovery Perception | Stage 2 - 10 minutes after endurance test in all tools
  The perception of recovery of the dominant lower limb will be evaluated through the Likert Scale of Recovery Perception, which consists of a scale with values between 1 and 10 points, 1 corresponding to no recovery and 10 to fully recovered
Participation of the anaerobic parameter | Stage 3 - During endurance test, until 7 minutes after test
  The total participation of the anaerobic parameter (PANA) will be calculated by the sum of the lactary anaerobic (CLAC) and alactic (CALA) contributions, analyzed by [lac] and the excess of post-exercise oxygen consumption (EPOC), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Marcelo Pastre, PhD, Study Director — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- State University of são Paulo, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No